CLINICAL TRIAL: NCT07175831
Title: Effect of Different Types of Exercise Intensities on Peak BDNF Oscillation Duration
Brief Title: Determination of BDNF Peak Time in Different Types of Exercises
Acronym: BDNF Kinematic
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aksaray University Training and Research Hospital (Other)
Responsible Party: Principal Investigator, serkan pancar, Assoc. Prof., Aksaray University Training and Research Hospital
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 30.06/07.10; Ethics Committe (Other: OKAT GAZİOSMANPAŞA UNIVERSITY RECTORATE/Social and Human Sciences Research Ethics Committee)
Record Dates: First submitted 2025-09-09; First posted 2025-09-16 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: BDNF; Lactate; Exercise Intensity; Healthy
Keywords: BDNF; Peak Time; Exercise Intensity
MeSH Terms: interventions — High-Intensity Interval Training

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Low-Intensity Continuous Training Group (n=4) (Experimental)
  Interventions: Behavioral: Low-Intensity Continuous Training
- Modarate-Intensity Interval Training Group (n=4) (Experimental)
  Interventions: Behavioral: Moderate intensity Interval training
- High-Intensity Interval Training Group (n=4) (Experimental)
  Interventions: Behavioral: High-Intensity Interval Training

INTERVENTIONS:
Behavioral: Low-Intensity Continuous Training — Participants ran continuously for 30 minutes at 50% of their MAS without rest.
  Other Names: LICE
  Arms: Low-Intensity Continuous Training Group (n=4)
Behavioral: Moderate intensity Interval training — Participants ran continuously for 30 minutes at 70% of their MAS without rest.
  Other Names: MICE
  Arms: Modarate-Intensity Interval Training Group (n=4)
Behavioral: High-Intensity Interval Training — Participants ran at 105-110% of their MAS for 15-second intervals, covering a pre-calculated distance during each bout. After each 15-second sprint, they rested passively for 15 seconds and returned to their starting point. This was repeated continuously for 5 minutes, constituting one set. A total of four 5-minute sets were completed, interspersed with 2,5-minute passive rest periods, yielding a total exercise time of 30 minutes.
  Other Names: HIIE
  Arms: High-Intensity Interval Training Group (n=4)

SUMMARY:
Purpose The purpose of this study was to determine the peak point of BDNF following exercises of different intensities.

Method This randomized crossover controlled trial aimed to examine the acute effects of three experimental conditions-high-intensity interval training, long-interval continuous training, and low-intensity continuous training-on serum BDNF and blood lactate levels in healthy young adults aged 18-25 years.

All participants completed the three conditions in a randomized and counterbalanced manner. To ensure balanced exposure, they were assigned to one of three groups (n = 4 per group), each following a distinct condition order based on a Latin square design. This approach guaranteed that each session occurred equally across time points (sessions 1-3) and that the order minimized sequence effects by rotating the position of each condition relative to the others.

To control for potential carryover-particularly from elevated neurochemical responses following intense exercise (BDNF increases had been reported)-no two high-intensity sessions were scheduled consecutively. Where possible, higher- and lower-intensity protocols were alternated. Furthermore, a seven-day interval separated each session to reduce residual physiological or cognitive effects.

The trial protocol was developed in line with CONSORT and SPIRIT guidelines, including relevant extensions for within-subject designs and non-pharmacological interventions. Participants were blinded to the study hypothesis.

All exercise sessions were conducted in the morning (09:00-11:00) on a track and field pitch under the supervision of a certified strength and conditioning coach to ensure consistency and adherence to protocol. Participants were instructed to avoid strenuous activity for 48 hours prior, abstain from alcohol and caffeine for 24 hours, and obtain at least 7-8 hours of sleep before each session. Dietary habits and general lifestyle were kept unchanged throughout the study.

During the first visit, participants' body weight and body fat percentage were assessed using bioelectrical impedance analysis. Resting heart rate was then recorded, followed by administration of the Yo-Yo Intermittent Recovery Test Level 1 to determine maximal aerobic speed (MAS), aerobic capacity, and peak heart rate.

In the following four visits, each participant completed all experimental conditions. Each exercise session began with a standardized 10-minute warm-up, including light jogging, dynamic stretching, and movement preparation drills.

All exercise sessions were conducted on a standard track and field facility and lasted 40 minutes in total, consisting of a 10-minute standardized warm-up, 24 minutes of exercise, and a 5-minute recovery period. The exercise component was individually prescribed based on each participant's MAS, determined from the Yo-Yo Intermittent Recovery Test Level 1. All running distances were calculated individually using time × speed formulas based on each participant's MAS, ensuring workload equivalence across conditions.

High-intensity interval exercise (HIIE): Participants ran at 105-110% of their MAS for 15-second intervals, covering a pre-calculated distance during each bout. After each 15-second sprint, they rested passively for 15 seconds and returned to their starting point. This was repeated continuously for 5 minutes, constituting one set. A total of four 5-minute sets were completed, interspersed with 2,5-minute passive rest periods, yielding a total exercise time of 30 minutes.

Moderate-Intensity Continuous Exercise (MICE): Participants ran continuously for 30 minutes at 70% of their MAS without rest.

Low-Intensity Continuous Exercise (LICE): Participants ran continuously for 30 minutes at 50% of their MAS without rest.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18 and 25 years
* No known medical condition that prevents participation in exercise
* Not currently using any pharmacological agents

Exclusion Criteria:

* Experiencing any discomfort before, during, or after exercise
* Current or past diagnosis of pharmacological or doping substance use
* Engaging in regular exercise (more than 3 times per week) within the last 2 weeks
* History of alcohol or substance addiction
* Any other condition or factor that may prevent full participation in the study protocol

Ages: 18 Years to 25 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Only male participants are eligible to participate in this study based on biological sex.
Enrollment: 12 (Actual)
Dates: Start 2025-05-10 (Actual); Primary Completion 2025-05-20 (Actual); Study Completion 2025-07-25 (Actual)

PRIMARY OUTCOMES:
BDNF | • Baseline, Immediately After Exercise (Day 1), 5 minute After Exercise (Day 1), 15 minutes After Exercise (Day 1), 30 minutes After Exercise (Day 1), 45 minutes After Exercise (Day 1), and 60 minutes After Exercise (Day 1).
  BDNF levels were measured using a Sunred brand ELISA kit from blood samples taken baseline and after exercise, and the results were reported in ng/mL units.
Lactate | • Baseline, Immediately After Exercise (Day 1), 5 minute After Exercise (Day 1), 15 minutes After Exercise (Day 1), 30 minutes After Exercise (Day 1), 45 minutes After Exercise (Day 1), and 60 minutes After Exercise (Day 1).
  Lactate levels were measured in millimoles per liter (mmol/L) from capillary/venous blood samples taken before and after exercise using a lactate analyzer.

CONTACTS AND LOCATIONS:
Locations (1):
- Aksaray university, Aksaray, Aksaray, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Birinci YZ, Pancar S, Simsek H, Soylu Y, Konuk K, Sahin S. Time-dependent comparison of serum BDNF responses following high-intensity interval exercise and moderate- and low-intensity continuous exercise in healthy young men. Sci Rep. 2026 Jan 31. doi: 10.1038/s41598-026-37728-z. Online ahead of print. PMID 41620464